CLINICAL TRIAL: NCT01439399
Title: Analgesic Efficacy of Intravenous Perfusion of Lidocaine, Ketamine or a Combination After Laparotomy in a Placebo-controlled, Randomized, Double-blind Prospective Study
Brief Title: Analgesic Efficacy of Intravenous Lidocaine and/or Ketamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Joray Florence, Chief Resident, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL-48h; 179/05 (Other: Cantonal Ethics Committee of Research on human)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; postoperative care; intravenous lidocaine; intravenous ketamine; morphine consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lidocaine (Active Comparator): Intravenous lidocaine administered preoperatively (anesthesia induction) and postoperatively during 48 hours
  Interventions: Drug: Lidocaine,
- Ketamine (Active Comparator): Intravenous ketamine administered preoperatively (anesthesia induction) and postoperatively during 48 hours
  Interventions: Drug: Ketamine
- Ketamine-Lidocaine (Active Comparator): Intravenous association of ketamine and lidocaine administered preoperatively (at anesthesia induction) and postoperatively during 48 hours.
  Interventions: Drug: association ketamine-lidocaine
- Saline 0,9% (Placebo Comparator): Control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine, — Lidocaine group received an IV bolus of 1.5 mg.kg-1 followed by a continuous infusion of 2 mg.kg-1.h-1 intraoperative and 1.33 mg.kg-1.h-1 for 48 h postoperative.
  Arms: Lidocaine
Drug: Ketamine — Ketamine group received a bolus of 0.5 mg.kg-1, then 0.25 mg.kg-1.h-1 followed by 0.1 mg.kg-1.h-1 for the first 24 h, then 0.05 mg.kg-1.h-1 for the next 24 h.
  Arms: Ketamine
Drug: association ketamine-lidocaine — Ketamine-lidocaine group received a bolus of 1.5 mg.kg-1 of lidocaine and 0.5 mg.kg-1 of ketamine, a continuous infusion of 1.3 mg.kg-1.h-1 of lidocaine and 0.17 mg.kg-1.h-1 of ketamine was delivered followed by 0.9 mg.kg-1 of lidocaine with 0.08 mg.kg-1.h-1 of ketamine during 48 h, the dose of ketamine being reduced to 0.04 mg.kg-1.h-1 after the first 24 hours.
  Arms: Ketamine-Lidocaine
Drug: Placebo — The control group (C) received an equal volume of saline 0.9 % during 48 h.
  Arms: Saline 0,9%

SUMMARY:
The aim of the present study is to evaluate the analgesic benefit of intravenous lidocaine and ketamine in the perioperative period of abdominal surgery.

DETAILED DESCRIPTION:
Optimal postoperative pain management facilitates rehabilitation immediately after abdominal surgery. Multiple studies have demonstrated that successful postoperative analgesia also reduces perioperative complications and improves patient comfort, thereby providing many benefits for the patient. In acute postoperative pain management intravenous lidocaine and/or ketamine have been advocated because of their morphine-sparing effect.

ELIGIBILITY:
Inclusion Criteria:

* abdominal surgery by laparotomy

Exclusion Criteria:

* laparoscopy
* history of chronic pain
* opioid self-administration
* psychiatric disorders
* difficulties with communication
* renal or hepatic dysfunction
* ASA physical status > 3

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine consumption | 48 hours
  Cumulative morphine consumption over 48 hours postoperatively

SECONDARY OUTCOMES:
Pain scores | 48 hours
  Pain scores at rest and movement
Mechanical hyperalgesia | 48 hours
  Mechanical hyperalgesia using pressure algometry
Occurrence of side effects | 48 hours
  Occurrence of side effects: sedation, nausea, vomiting, itching, nightmares

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kern, Study Director — University of Lausanne Hospitals
Locations (1):
- University Hospital Center and University, Lausanne, Canton of Vaud, Switzerland